CLINICAL TRIAL: NCT01247116
Title: First-line Bosentan and Sildenafil Combination Therapy for Pulmonary Arterial Hypertension: A Safety and Efficacy Pilot Study
Brief Title: First-line Bosentan and Sildenafil Combination Therapy for Pulmonary Arterial Hypertension
Status: Completed | Type: Observational
Sponsor: University of Calgary (Other)
Collaborators: Actelion (Industry)
Responsible Party: Principal Investigator, Naushad Hirani, Clinical Assistant Professor, University of Calgary
Other Study IDs: BSC-UOC-2009
Record Dates: First submitted 2010-11-23; First posted 2010-11-24 (Estimated); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Hypertension, Pulmonary
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate the strategy of initiating double oral combination therapy with bosentan and sildenafil at the time of diagnosis of pulmonary arterial hypertension (PAH) in a preliminary way.

DETAILED DESCRIPTION:
Current treatment paradigms for PAH suggest adopting goals of therapy with relatively objective parameters such as 6 minute walk distance to determine when to add a second oral agent (1). This often entails observing deterioration in the patient on a single agent before instituting the second one. This strategy could be problematic, as patients may never recover the function lost due to progressive PAH (2). In addition, given the malignant nature of the clinical course of PAH in many cases and the nature of the underlying proliferative vasculopathy, some have argued that altering this paradigm to resemble that used in cancer chemotherapy may be more appropriate (3). That is, "induction" therapy at diagnosis with multiple agents followed by a maintenance phase of treatment might offer significant benefits to the patient.

This open-label pilot study is the first to investigate the potential efficacy and safety of a first-line combination strategy in consecutive patients with PAH in contrast to the "add-on" strategy for combination therapy. It will serve as the basis on which to consider larger, multicenter investigations of this strategy.

1. Hoeper M, et al. Eur Respir J. 2005 Nov;26(5):858-63.
2. Halpern SD, et al. Proc Am Thorac Soc. 2008 Jul 15;5(5):631-5.
3. Provencher S, et al. Chest. 2005 Dec;128(6 Suppl):622S-628S.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic Functional Class III PAH in the following categories: Idiopathic (IPAH), Familial (FPAH), Associated with connective tissue disease, Associated with drugs or toxins
* PAH diagnosed by right heart catheterization, defined as: mean pulmonary arterial pressure (mPAP) ≥ 25 mmHg, PVR > 3 mmHg/l/min (Wood units) or > 240 dyn sec cm-5, pulmonary capillary wedge pressure (PCWP) ≤ 15 mmHg
* Baseline 6 MWT distance > 150 and < 450 m

Exclusion Criteria:

* Treatment with ERAs other than bosentan;
* Treatment with PDE5 inhibitors other than sildenafil;
* Treatment with any prostanoid;
* PAH associated with thyroid disorders, glycogen storage disease, Gaucher disease, hereditary hemorrhagic telangiectasia, hemoglobinopathies, myeloproliferative disorders and splenectomy; valvular disease with valvular lesions to be excluded by echocardiogram within 2 years prior to randomization
* Restrictive lung disease: total lung capacity (TLC) < 60% of normal predicted value;
* Obstructive lung disease: forced expiratory volume/forced vital capacity (FEV1/FVC) < 50%

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with idiopathic pulmonary arterial hypertension (IPAH) or PAH associated with connective tissue disease that are naive to PAH targeted therapies will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2009-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
6 minute walk test distance | 4 months

SECONDARY OUTCOMES:
6 minute walk test distance | 12 months
Echocardiographic parameters | 4 months
Hemodynamics | 4 months
Quality of Life as measured by CAMPHOR questionnaire | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Naushad Hirani, MD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Peter Lougheed Hospital, Calgary, Alberta, Canada